CLINICAL TRIAL: NCT02003365
Title: An Open-label, Single Administration Study to Characterize the Local Duration of Exposure of Triamcinolone Acetonide From FX006 in Patients With Osteoarthritis (OA) of the Knee
Brief Title: Study to Characterize the Local Duration of Exposure From FX006 in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX006-2013-005
Record Dates: First submitted 2013-11-18; First posted 2013-12-06 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee; corticosteroids; triamcinolone acetonide; synovial fluid
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — FX006

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- FX006 10 mg (Experimental): Single 3 mL intra-articular (IA) injection
  Interventions: Drug: FX006 10 mg
- FX006 40 mg (Experimental): Single 3 mL intra-articular (IA) injection
  Interventions: Drug: FX006 40 mg
- TCA IR 40 mg (Active Comparator): Single 1 mL intra-articular (IA) injection
  Interventions: Drug: TCA IR 40 mg

INTERVENTIONS:
Drug: FX006 10 mg — Extended-release formulation
  Arms: FX006 10 mg
Drug: FX006 40 mg — Extended-release formulation
  Arms: FX006 40 mg
Drug: TCA IR 40 mg — Immediate-release formulation
  Other Names: Kenalog®-40 Injection; Triamcinolone Acetonide Crystalline Suspension (TAcs)
  Arms: TCA IR 40 mg

SUMMARY:
The purpose of this study was to characterize the local duration of exposure of TCA for 2 doses of FX006 relative to 40 mg of TCA IR in patients with OA of the knee.

DETAILED DESCRIPTION:
This study was an open-label, single administration design, conducted in male and female patients ≥40 years of age with OA of the knee.

Patients were enrolled sequentially with 8 patients per cohort, as follows:

Cohort A: FX006 40 mg, Final Visit at Week 20 Cohort B: FX006 40 mg, Final Visit at Week 16 Cohort C: FX006 10 mg, Final Visit at Week 12 Cohort D: FX006 40 mg, Final Visit at Week 12 Cohort E: Triamcinolone acetonide immediate-release (TCA IR) 40 mg, Final Visit Week 12

Each patient was evaluated for up to 12, 16, or 20 weeks following a single IA injection depending on the assigned cohort. Following the screening visit, safety was evaluated at 3 out-patient visits and synovial fluid was collected at Day 1 for baseline measurements and the Final Visit for drug concentration measurements.

ELIGIBILITY:
Key Inclusion Criteria:

* Written consent to participate in the study
* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Has documented diagnosis of OA of the index knee made at least 6 months prior to Screening
* Currently meets American Collage of Rheumatology Criteria (clinical and radiological) for OA
* Index knee pain for >15 days over the last month
* Body mass index (BMI) ≤ 40 kg/m2
* Ambulatory and in good general health

Key Exclusion Criteria:

* History of Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis or amyloidosis
* History of arthritides due to crystals (e.g., gout, pseudogout)
* History of infection in the index joint
* Clinical signs and symptoms of active knee infection or crystal disease of the index knee
* Presence of surgical hardware or other foreign body in the index knee
* Unstable joint (such as a torn anterior cruciate ligament) within 12 months of Screening
* IA corticosteroid (investigational or marketed) in any joint within 6 months of Screening
* IA hyaluronic acid (investigational or marketed) in the index knee within 6 months of Screening
* Oral corticosteroids (investigational or marketed) within 1 month of Screening
* Inhaled, intranasal and topical corticosteroids (investigational or marketed) within 2 weeks of Screening
* Any other IA investigational drug/biologic within 6 months of Screening
* Prior use of FX006
* Prior arthroscopic or open surgery of the index knee within 12 months of Screening
* Planned/anticipated surgery of the index knee during the study period
* Active or history of malignancy within the last 5 years, with the exception of resected basal cell carcinoma, squamous cell carcinoma of the skin, or resected cervical atypia or carcinoma in situ

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bodick, MD, Study Director — Flexion Therapeutics
Locations (3):
- United States (3):
  - Paducah, Kentucky
  - Duncansville, Pennsylvania
  - Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study took place at 3 centers across the United States. Enrollment took approximately 2 months.
Pre-assignment Details: Subjects were screened for eligibility within 14 days of being enrolled
Groups:
- FX006 10 mg: 10 subjects received FX006 10 mg as a single 3 mL IA injection
- FX006 40 mg: 30 Subjects received FX006 40 mg as a single 3 mL IA injection
- TCA IR 40 mg: 10 subjects received TCA IR 40 mg as a single 1 mL IA injection
Period: Overall Study
Arm/Group | FX006 10 mg | FX006 40 mg | TCA IR 40 mg
Started | 10 | 30 | 10
Completed | 10 | 30 | 9
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FX006 10 mg; FX006 40 mg: Single 3 mL IA injection
- TCA IR 40 mg: Single 1 mL IA injection
- Total: Total of all reporting groups
Arm/Group | FX006 10 mg | FX006 40 mg | TCA IR 40 mg | Total
Number analyzed (Participants) | 10 | 30 | 10 | 50
Age, Continuous [Mean (Full Range); unit: years] | 61.5 [49 to 69] | 62.8 [48 to 78] | 61.6 [52 to 75] | 62.15 [48 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 20 | 7 | 34
  Male | 3 | 10 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Triamcinolone Acetonide in Synovial Fluid
Description: Analyses of synovial fluid drug concentrations were performed using the Synovial Fluid Drug Concentration Population.
  Values recorded as lower limit of quantification (LLOQ) (< 50 pg/mL) were counted as half the value below limit of quantification (BLQ).
Time Frame: 12 to 20 weeks
Population: All patients who received study drug and had synovial fluid obtained at the Final Visit were included in the Synovial Fluid Drug Concentration Population.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | FX006 10 mg | FX006 40 mg | TCA IR 40 mg
Number analyzed (Participants) | 8 | 15 | 5
pg/mL
  Week 12 | 477.5 [166.41 to 1369.91] | 923.7 [74.24 to 11492.46] | 250.1 [0.16 to 380930.9]
  Week 16 | NA [NA to NA] — For the 10 mg group of FX006 patients were only followed until week 12. | 224.3 [37.42 to 1344.70] | NA [NA to NA] — TCA IR 40 mg group patients were only followed until week 12.
  Week 20 | NA [NA to NA] — For the 10 mg group of FX006 patients were only followed until week 12. | 33.3 [20.28 to 54.74] | NA [NA to NA] — TCA IR 40 mg group patients were only followed until week 12.

2. Secondary Outcome: Plasma Drug Concentrations by Time
Description: Plasma Drug Concentration Population. Analyses of plasma drug concentrations were performed using the Plasma Drug Concentration Population.
  Values recorded as lower limit of quantification (LLOQ) (< 10 pg/mL) were counted as half the value below limit of quantification (BLQ).
Time Frame: Weeks 6, 12, 16 and 20
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | FX006 10 mg | FX006 40 mg | TCA IR 40 mg
Number analyzed (Participants) | 10 | 30 | 10
pg/mL
  Week 6 | 26.5 [15.09 to 46.59] | 100.1 [76.05 to 131.80] | 21.1 [5.76 to 77.13]
  Week 12 | 6.6 [4.26 to 10.26] | 8.9 [3.97 to 19.79] | 9.4 [1.86 to 47.40]
  Week 16 | NA [NA to NA] — For the 10 mg group of FX006 patients were only followed until week 12. | 26.4 [8.75 to 79.64] | NA [NA to NA] — For the TCA IR 40 mg group patients were only followed until week 12.
  Week 20 | NA [NA to NA] — For the 10 mg group of FX006 patients were only followed until week 12. | 10.1 [4.21 to 24.48] | NA [NA to NA] — For the TCA IR 40 mg group patients were only followed until week 12.

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored/assessed from post-injection on Day 1 through 12 weeks for FX006 10 mg and TCA IR groups and up to 20 weeks for FX006 40 mg groups.
Groups:
- TCA IR: Single 1 mL IA injection
Arm/Group | FX006 10 mg | FX006 40 mg | TCA IR
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/30 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/30 | 2/10
Other Adverse Events (participants affected / at risk) | 5/10 | 5/30 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 10 mg (N=10) | FX006 40 mg (N=30) | TCA IR (N=10)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Food Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 10 mg (N=10) | FX006 40 mg (N=30) | TCA IR (N=10)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Food Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Frostbite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes